CLINICAL TRIAL: NCT02170311
Title: "Phase Ib Study of Z-213 in Subjects With Iron-deficiency Anemia - To Investigate the Safety, Tolerability Pharmacokinetics and Pharmacodynamics -"
Brief Title: Pharmacokinetics, Pharmacodynamics and Safety Study of Z-213 to Iron Deficiency Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Z213-01
Record Dates: First submitted 2014-06-10; First posted 2014-06-23 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Iron Deficiency Anemia
Keywords: Z-213, Ferric carboxymaltose, Iron, Iron-deficiency-anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Z-213 100mg (Experimental): Group/Cohort Label: 100 mg iron Z-213 will be administered by intravenous infusion.
  Interventions: Drug: Z-213
- Z-213 500mg (Experimental): Group/Cohort Label: 500 mg iron Z-213 will be administered by intravenous infusion.
  Interventions: Drug: Z-213
- Z-213 800mg (Experimental): Group/Cohort Label: 800 mg iron Z-213 will be administered by intravenous infusion.
  Interventions: Drug: Z-213
- Z-213 1000mg (Experimental): Group/Cohort Label: 1000 mg iron Z-213 will be administered by intravenous infusion.
  Interventions: Drug: Z-213

INTERVENTIONS:
Drug: Z-213

SUMMARY:
The safety, tolerability, pharmacokinetics and pharmacodynamics of Z-213 will be investigated in patients with iron-deficiency anemia after administration of a single dose (100 mg, 500 mg, 800 mg or 1,000 mg iron).

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild iron deficiency anemia

Exclusion Criteria:

* Patients with anemia caused by conditions other than iron deficiency
* Patients with abnormal laboratory test values at screening for C-reactive protein, Serum phosphorus, Aspartate aminotransferase, Alanine aminotransferase, Total bilirubin
* Patients with liver, kidney or circulatory system disease
* Patients with a history or present illness that is a malignant tumor or autoimmune disease
* Patients who underwent intravenous administration of an iron preparation, administration of an erythropoiesis stimulation agent or blood transfusion within 8 weeks before the screening
* Patients who underwent oral administration of an iron preparation (including an over-the-counter drug or supplement) within 4 weeks before the screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of total serum iron (Cmax), (Tmax), (AUC0-t), (AUC0-24),(AUC0-72),(T1/2), (CL), (Vd, area), (Vd, ss), (MRT) or total urine iron (CLren), (Ae). | 8days

CONTACTS AND LOCATIONS:
Overall Officials: Zeria Investigator, Study Director — Zeria Pharmaceutical Co., Ltd
Locations (1):
- Zeria Investigative Site, Tokyo, Japan